CLINICAL TRIAL: NCT01328912
Title: Remote Ischemic Preconditioning in High Risk Cardiovascular Surgery Patients: A Randomized Controlled Trial
Brief Title: Remote Ischemic Preconditioning in High Risk Cardiovascular Surgery Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Darrin Payne, MD, MSC, BSc, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6576
Record Dates: First submitted 2011-03-31; First posted 2011-04-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Death; Stroke; Low Cardiac Output Syndrome; Myocardial Infarction; Renal Failure; Pulmonary Failure
Keywords: ischemic preconditioning; cardiac surgery; vascular surgery
MeSH Terms: conditions — Death; Stroke; Cardiac Output, Low; Myocardial Infarction; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote ischemic preconditioning stimulus (Experimental)
  Interventions: Other: Remote ischemic preconditioning stimulus
- Control (Placebo Comparator)
  Interventions: Other: control

INTERVENTIONS:
Other: Remote ischemic preconditioning stimulus — The intervention will consist of 3 cycles of 5 minutes of upper limb ischemia. The RIPC stimulus will be performed using a blood pressure cuff placed on the upper arm inflated above systemic pressure to 200 mmHg for 5 minutes, then deflated for 5 minutes. Ischemia will be assured with the use of a saturation probe on the digit of the involved arm.
  Arms: Remote ischemic preconditioning stimulus
Other: control — These patients are randomized to placebo, thus they will no undergo the RIPC stimulus.
  Arms: Control

SUMMARY:
Remote ischemic preconditioning (RIPC) occurs when a tissue (ex. heart) becomes less vulnerable to an ischemic insult if a remote tissue (ex. arm) has had previous exposure to a period of ischemia and reperfusion. A beneficial effect of RIPC has been demonstrated in several randomized studies in patients undergoing cardiac and vascular surgery, as well as interventional cardiac procedures such as angioplasty. They have shown improvements in cardiac, renal, neurologic and respiratory function. Most have focused on surrogate outcomes, such as biochemical markers of cardiac and renal function in low-risk patients. No trials have investigated only high-risk patients or been designed to detect clinical outcomes.

This study is a randomized-controlled trial powered to detect clinical events in a high-risk cohort undergoing cardiovascular surgery. Patients will be randomized to RIPC (exposed to cycles of inflation of a blood pressure cuff on the upper arm prior to undergoing surgery) or control (no ischemic stimulus).

The investigators hypothesize this population will demonstrate lower rates of adverse ischemic events. The investigators also intend to sample biochemical markers to better elucidate the mechanism of RIPC and generate hypotheses for future studies and interventions. Post-operatively the investigators will monitor for adverse clinical outcomes including cardiac, renal, pulmonary and neurologic injury.

RIPC is simple, inexpensive and easily reproducible and there have been no reports of adverse consequences. Post-operative ischemic events such as stroke, myocardial infarction, cardiac, renal and respiratory failure affect patient survival and quality of life, and represent a sizeable financial burden to health care. If beneficial effects of RIPC are demonstrated, it will be widely applicable to the entire population of cardiac and vascular patients resulting in a widely-implemented change in practice.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing either cardiac or vascular surgical procedures and are deemed to be at increased risk of suffering adverse ischemia-related events (judged by pre-operative evidence of clinical ischemic conditions, pre-operative screening indicating cardiovascular disease or undergoing higher-risk surgery).

Exclusion Criteria:

* Will not include emergency cases, patients with known vascular disease (ex. arterial occlusive disease, arterio-venous shunts) or neurologic disease affecting the upper limb and patients unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2012-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be a composite of clinical MACE (Multiple Adverse Cardiovascular Events), incorporating all-cause mortality, myocardial infarction, stroke, respiratory failure, acute renal failure and low cardiac output syndrome | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Darrin Payne, MD, Principal Investigator — Queen's University / Kingston General Hospital
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada